CLINICAL TRIAL: NCT03218267
Title: Does the Total Hip Replacement Impact of Postural Stability?
Brief Title: The Postural Control in Patients After Total Hip Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Małgorzata Eliks, Assistant, MSc, Poznan University of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 949/14
Record Dates: First submitted 2017-07-10; First posted 2017-07-14 (Actual); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Total Hip Replacement
Keywords: total hip replacement; static disbalance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individuals after total hip replacement (Experimental): Individuals after total hip replacement. Patients treated at the Out-Patient Ward of W. Dega Orthopaedic-Rehabilitation Clinical Hospital of Karol Marcinkowski University of Medical Sciences in Poznań. The examination of participants included the static posturography and one-leg standing test.
  Interventions: Other: Static Posturography; Other: One-leg standing test (OLS)
- control group (Active Comparator): The group with healthy individuals; without total hip replacement. The examination of participants included the static posturography and one-leg standing test.
  Interventions: Other: Static Posturography; Other: One-leg standing test (OLS)

INTERVENTIONS:
Other: Static Posturography — The balance platform (Good Balance by Metitur) and one leg standing test (OLS) were used to assess the static balance. OLS test was performed on left and right foot separately. The static posturography was performed with several various positions of feet. Position : normal standing with eyes open and eyes closed - an upright standing with feet placed parallel 20 cm apart for 30 s. Position: tandem - a stance with one foot placed ahead of the other for 10 s. Position: second form of tandem - a stance with one foot placed ahead of the other with feet placed on both sides of the line dividing platform to two parts for 20s. Position: one leg standing: stance on the one leg for 5 s.
Other: One-leg standing test (OLS) — During the one-leg standing test (OLS) the time of maintain this position by the patients was measured. The placement of the limbs was the same as in the case of the balance platform test. Subjects performed 3 trials on each lower limb. Time ended when subject either: loosed balance and touched raised foot the floor, moved supporting leg on the ground, a significant loss of balance or a maximum of 60 s had elapsed. Results achieved by the subjects after THR on both operated (OLS-O) and non operated limbs (OLS-N) were compared with the index of the control group (OLS-C: mean result of the tests performed on the left and right legs).

SUMMARY:
Total hip replacement (THR) is the procedure which can improve the quality of life in patients with osteoarthritis. However, deficits in static stability and impairment of the lower limb efficiency can be observed even several months after procedure. The aim of this study was to investigate the static balance of the standing position in patients treated by THR.

DETAILED DESCRIPTION:
The balance platform and one leg standing test (OLS) were used to assess the static balance. The postural balance tests were performed on the Metitur Good Balance platform. Static balance tests on balance platform were performed in several position with different foot placement like: normal standing with eyes open (NS EO) and eyes closed (NS EC) position, tandem position (TP), second form of tandem position (2TP) and one leg standing position (1L). Participants were asked to maintain the motionless upright position with both arms at their sides and eyes staring at a target in front of them.

During the normal standing (NS) position the patient stood on the platform barefoot with the feet placed parallelly (symmetric position of feet) with a 20 cm distance between them. The length of the trials with EO and EC was 30 seconds each.

In TP (tandem position) the width of base of support was narrowed down significantly, therefore test lasted only 10 s. During the test in TP one foot was placed directly in the front of the other (on the line) and the heel of the front foot was touched the toes of the rear foot. Tests were performed tests in TP with the left foot in front (TLF) and with right foot in front (TRF) separately. In THR group the placement of the operated limb in the front stance was called the TOF test, while the placement of the non operated limb in the front stance was called the TNF test. The results obtained in TOF position and TNF position were compared with tandem control index (TC - mean of results obtained from control group in TLF and TRF positions).

In 2TP alternately left or right foot was places in front of the other, but the feet were placed on both sides of the line dividing platform to two parts (line was tangent to the medial edge of feet). The length of exercise was 20 s. Analogically to the tandem test, patients were examined with the operated (2TOF) and non operated limb (2 TNF) in the front. Results were compared to the second tandem control index (2TC) representing the mean results of the control group as was described above.

When testing one leg standing position on the balance platform, the patients were asked to raise one foot half the level of the calf of the supporting leg but not touching the stance limb. The trial lasted for 5 s. The test was stopped when the subject used his arms (touched the handrail) or used the raised foot (touched the floor). Usually after 2 failed attempts or fear of falling down procedure was stopped and results was not recording. The results of the patients after THR when standing on the operated (1 O) and non operated (1 N) leg were compared to the index denoting the mean results of the control group (1 C).

During the static tests we analyzed the mean velocity of sway of the center of feet pressure (COP) in the frontal plane (X, mm/s) and in the sagittal plane (Y, mm/s) and the value of the middle of spectrum in the same planes. The spectrum is characterised by two co-dependent variables such as frequency (Hz) and the excursion (mm).

During the one-leg standing test (OLS) the time of maintain this position by the patients was measured. The placement of the limbs was the same as in the case of the balance platform test. Subjects performed 3 trials on each lower limb. Time ended when subject either: loosed balance and touched raised foot the floor, moved supporting leg on the ground, a significant loss of balance or a maximum of 60 s had elapsed. Results achieved by the subjects after THR on both operated (OLS-O) and non operated limbs (OLS-N) were compared with the index of the control group (OLS-C: mean result of the tests performed on the left and right legs).

ELIGIBILITY:
Inclusion Criteria:

* for patients: total hip replacement the minimum of 6 months period since the procedure, age above 55 years, unassisted gait, and the minimum of 9 points on the AMTS scale
* for healthy volunteers: without total hip replacement age above 55 years, unassisted gait, and the minimum of 9 points on the AMTS scale

Exclusion Criteria:

* for patients: neurological diseases, muscles diseases, rheumatic diseases (rheumatoid arthritis, ankylosing spondylitis, psoriatic arthritis) and sciatica. Additionally we excluded patients who had operations in the area of the spine and lower limbs (knee arthroscopy with ACL reconstruction or meniscectomy, total knee replacement, total hip replacement in both extremities, osteotomy or arthrodesis).
* for healthy volunteers: neurological diseases, muscles diseases, rheumatic diseases (rheumatoid arthritis, ankylosing spondylitis, psoriatic arthritis) and sciatica. Additionally we excluded patients who had operations in the area of the spine and lower limbs (knee arthroscopy with ACL reconstruction or meniscectomy, total knee replacement, total hip replacement in both extremities, osteotomy or arthrodesis).

Ages: 59 Years to 83 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2015-09-01 (Actual); Study Completion 2016-05-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of mean COP velocity in anteroposterior and mediolateral directions during stance in subjects. | 6 months
  Mean COP velocity [mm/s] and the value of the middle of spectrum [Hz; mm] is recorded in anteroposterior (AP) and mediolateral (ML) directions within posturographic evaluation in examination of every participant
  Evaluation of mean COP velocity in anteroposterior and mediolateral directions during stance in subjects. Mean COP velocity [mm/s] and the value of the middle of spectrum [Hz; mm] is recorded in anteroposterior (AP) and mediolateral (ML) directions within posturographic evaluation in examination of every participant

SECONDARY OUTCOMES:
Evaluation of the time of maintain one-leg standing position by the patients. | 6 months
  The time of maintain one-leg standing position on each limb is assessed in every participants.
  The result is expressed in seconds [s]. The time of maintain one-leg standing position on each limb is assessed in every participants.
  The result is expressed in seconds [s].

CONTACTS AND LOCATIONS:
Overall Officials: Przemysław Lisiński, PhD, Prof., Study Director — Poznan University of Medical Sciences; Agnieszka Wareńćzak, PhD, Principal Investigator — Poznan University of Medical Sciences

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wykman A, Goldie I. Postural stability after total hip replacement. Int Orthop. 1989;13(4):235-8. doi: 10.1007/BF00268504. PMID 2599698
- [Background] Nantel J, Termoz N, Ganapathi M, Vendittoli PA, Lavigne M, Prince F. Postural balance during quiet standing in patients with total hip arthroplasty with large diameter femoral head and surface replacement arthroplasty. Arch Phys Med Rehabil. 2009 Sep;90(9):1607-12. doi: 10.1016/j.apmr.2009.01.033. PMID 19735790
- [Background] Calo L, Rabini A, Picciotti PM, Laurino S, Passali GC, Ferrara PE, Maggi L, Piazzini DB, Specchia A, Frasca G, Ronconi G, Bertolini C, Scarano E. Postural control in patients with total hip replacement. Eur J Phys Rehabil Med. 2009 Sep;45(3):327-34. Epub 2009 Feb 11. PMID 19209135
- [Background] Springer BA, Marin R, Cyhan T, Roberts H, Gill NW. Normative values for the unipedal stance test with eyes open and closed. J Geriatr Phys Ther. 2007;30(1):8-15. doi: 10.1519/00139143-200704000-00003. PMID 19839175
- [Background] Lui RC, Johnson FE, Horovitz JH, Cunningham JN Jr. Aortoesophageal fistula: case report and literature review. J Vasc Surg. 1987 Oct;6(4):379-82. doi: 10.1067/mva.1987.avs0060379. PMID 3309380
- [Background] Balogun JA, Ajayi LO, Alawale F. Determinants of single limb stance balance performance. Afr J Med Med Sci. 1997 Sep-Dec;26(3-4):153-7. PMID 10456159
- [Background] Truszczynska A, Drzal-Grabiec J, Rapala K, Gmitrzykowska E. Postural stability in patients with osteoarthritis of the hip. Pilot study. Ortop Traumatol Rehabil. 2013 Nov-Dec;15(6):567-73. doi: 10.5604/15093492.1091512. PMID 24662903
- [Background] Rougier P, Belaid D, Cantalloube S, Lamotte D, Deschamps J. Quiet postural control of patients with total hip arthroplasty following joint arthritis. Motor Control. 2008 Apr;12(2):136-50. doi: 10.1123/mcj.12.2.136. PMID 18483448
- [Derived] Warenczak A, Lisinski P. Does total hip replacement impact on postural stability? BMC Musculoskelet Disord. 2019 May 17;20(1):229. doi: 10.1186/s12891-019-2598-9. PMID 31101048